CLINICAL TRIAL: NCT04492826
Title: Evaluation of the Occurrence of Postoperative Surgical Site Infection in Otolaryngology Flap Surgery With Bone Graft, a Retrospective Analytic Study Between 2012 and 2019
Brief Title: Postoperative Surgical Site Infection afterENT Bone Flap Surgery
Acronym: SSI-flap
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20_5052
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Rate of Infections; Operating Site; Post-operative Surgery; Bone Flap Surgery; Otolaryngology
Keywords: bone flap surgery; postoperative surgical infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infected patients: patients with bone flap surgeries
  Interventions: Procedure: Postoperative infections rate

INTERVENTIONS:
Procedure: Postoperative infections rate — Assess the postoperative infection rate after otolaryngology bone flap surgery.

SUMMARY:
In 2017, the French Society in anesthesia and reanimation published new recommendations on intraoperative antibiotic prophylaxis. Now, no more than 48 hours of antibiotic prophylaxis applies to any otolaryngology surgery, regardless of patient's medical history or type of flap used to rebuild. This has resulted in an alignment of our local protocol in Croix-Rousse hospital.

However, after few years, our local impressions are that bone flap surgeries are very likely to provide surgical site infections (osteo-articular or non-osteo-articular infections).

The prejudice of these postoperative site infections is significant, with serious consequences,. of both functional and aesthetic sides.

We wanted to objectify this impression by retrospectively analyzing the data relating to patients operated on for bone flapsurgeries.

Knowing the operation site infection rate after surgery for otolaryngology bone flap surgery will allow us to objectively understand the infectious risk of these surgeries, in particular the risk of osteoarticular infection. Identifying operation site infection factors will allow us to better target and prevent them.

The goal is to find out if the antibiotic prophylaxis currently recommended is sufficient and effective for this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated for bone flap in Croix-Rousse hospital, in otorhinolaryngology department, since september 2012 and until January 2019

Exclusion Criteria:

* patient's opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient operated on for bone flap surgery by the Otorhinolaryngology surgery team in Croix-Rousse hospital (Pr CERUSE)
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Postoperative infections rate after otolaryngology bone flap surgery | 1 year
  Assess the postoperative infection rate after bone flap otolaryngology surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France